CLINICAL TRIAL: NCT02939326
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Dose Cohort Study to Evaluate Safety and Efficacy of a Single Treatment Cycle of EB-001 in Subjects With Glabellar Frown Lines
Brief Title: Evaluate Safety and Efficacy of a Single Treatment Cycle of EB-001 in Subjects With Glabellar Frown Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bonti, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB001-GL201
Record Dates: First submitted 2016-10-11; First posted 2016-10-20 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Glabellar Frown Lines (GL)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- Placebo (Placebo Comparator): Intervention: Drug: Placebo
  Single Injection of placebo into five (5) 0.1 mL IM injections into glabellar area.
  Interventions: Drug: Placebo injection
- EB-001 Dose 1 (1X) (Active Comparator): Intervention: Drug: EB-001
  Single Injection of Low Dose of EB-001 into five (5) 0.1 mL IM Injections into glabellar area
  Interventions: Drug: EB-001 injection
- EB-001 Dose 2 (3X) (Active Comparator): Intervention: Drug: EB-001, 3X Dose 1
  Single Injection of EB-001 into five (5) 0.1 mL IM Injections into glabellar area
  Interventions: Drug: EB-001 injection
- EB-001 Dose 3 (9X) (Active Comparator): Intervention: Drug: EB-001, 9X Dose 1
  Single Injection of EB-001 into five (5) 0.1 mL IM Injections into glabellar area
  Interventions: Drug: EB-001 injection
- EB-001 Dose 4 (12X) (Active Comparator): Intervention: Drug: EB-001, 12X Dose 1
  Single Injection of EB-001 into five (5) 0.1 mL IM Injections into glabellar area
  Interventions: Drug: EB-001 injection
- EB-001 Dose 5 (16X) (Active Comparator): Intervention: Drug: EB-001, 16X Dose 1
  Single Injection of EB-001 into five (5) 0.1 mL IM Injections into glabellar area
  Interventions: Drug: EB-001 injection
- EB-001 Dose 6 (21X) (Active Comparator): Intervention: Drug: EB-001, 21X Dose 1 Single Injection of EB-001 into five (5) 0.1 mL IM Injections into glabellar area
  Interventions: Drug: EB-001 injection
- EB-001 Dose 7 (28X) (Active Comparator): Intervention: Drug: EB-001, 28X Dose 1
  Single Injection of Highest Dose of EB-001 into five (5) 0.1 mL IM Injections into glabellar area
  Interventions: Drug: EB-001 injection

INTERVENTIONS:
Drug: EB-001 injection
  Other Names: Botulinun Toxin Type E
  Arms: EB-001 Dose 1 (1X); EB-001 Dose 2 (3X); EB-001 Dose 3 (9X); EB-001 Dose 4 (12X); EB-001 Dose 5 (16X); EB-001 Dose 6 (21X); EB-001 Dose 7 (28X)
Drug: Placebo injection
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of EB-001 compared to placebo in subjects with glabellar frown lines (GL).

DETAILED DESCRIPTION:
This study of EB-001 to measure safety and efficacy in GL. Single doses of EB- 001 administered through IM injection into procerus at midline and the medial and lateral corrugators will be assessed in healthy subjects with glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated IRB-approved informed consent form (ICF).
2. Men or women between the ages of 18 and 60, inclusive.
3. Subjects in good health as determined by medical history, physical and focused neurological examinations, clinical laboratory studies, electrocardiograms (ECGs), vital signs, and Investigator's judgement.
4. Presence of bilaterally symmetrical GL of moderate to severe rating at maximum frown, as measured using FWS by both the Investigator and subject prior to study treatment.
5. Subjects with sufficient visual acuity without the use of eyeglasses (contact lens use acceptable) to accurately assess their facial wrinkles as determined by Investigator's judgement.
6. Women of child bearing potential must not be pregnant, lactating, or planning to become pregnant during the study.
7. Women of non-childbearing potential must be either postmenopausal (at least 12 consecutive months of amenorrhea) or surgically sterile (e.g., tubal ligation, hysterectomy, etc.).
8. Women of childbearing potential agreeing to use dual methods of contraception from the day of dosing until 3 months afterwards. Female subjects using oral contraception must have initiated treatment at least 2 months prior to the day of dosing.
9. Male subjects with partner(s) of childbearing potential agreeing to use dual methods of contraception from the day of dosing until 3 months afterwards, and to no sperm donation from day of dosing until 3 months afterwards.
10. Willing and able to complete protocol requirements and instructions, which include completion of all required visits.

Exclusion Criteria:

1. Any condition that precludes a subject's ability to comply with study requirements, including completion of the study visits or inability to read, understand, and/or self-assess GL severity using FWS.
2. Any uncontrolled systemic disease or other medical condition.
3. Any medical condition that may put the subject at increased risk with exposure to botulinum toxin of any serotype, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
4. Current or previous botulinum toxin treatment of any serotype.
5. Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study treatment).
6. Known immunization or hypersensitivity to any botulinum toxin serotype.
7. Known allergy or sensitivity to any of the components of the study treatments, or any materials used in the study procedures.
8. Any of the following procedures or treatments occurring within the specified period prior to screening:

   * 3 months: Non-ablative resurfacing laser or light treatment, microdermabrasion, or superficial peels.
   * 6 months: Any facial cosmetic procedure with medium depth to deep facial chemical peels (e.g., trichloroacetic acid [TCA] and phenol), or mid facial or periorbital laser skin resurfacing.
   * 6 months: On topical retinoid therapy and/or topical hormone cream applied to the face, who have not been on a consistent dose regimen and are unable to maintain the same regimen for the study.
   * 12 months: Mid-facial or periorbital treatment with non-permanent soft tissue fillers.
   * 12 months: On oral retinoid therapy.
9. Prior periorbital surgery, facial lift (full face or mid face), brow lift, or related procedures (e.g., eyelid [blepharoplasty] and/or eyebrow surgery).
10. Prior mid face or periorbital treatment with permanent soft tissue fillers, synthetic implantation (e.g., Gore-Tex®), and/or autologous fat transplantation.
11. Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin.
12. The inability to substantially lessen facial rhytides (fixed lines) even by physically spreading them apart, as determined by the Investigator.
13. Permanent make-up that would interfere with the assessment of facial wrinkles.
14. Subjects who, in the Investigator's opinion, are unable or unwilling to maintain their standardized skin care regimen throughout the study period.
15. Any eyebrow or eyelid ptosis at baseline as determined by the Investigator.
16. Infection or skin disorder at the injection sites.
17. History of facial nerve palsy.
18. Recent history (within 6 months of screening) of alcohol or drug abuse based on the Investigator's judgement.
19. Anticipated need for surgery or overnight hospitalization during the study. Current enrollment in an investigational drug or device study or participation in such a study within 30 days or 5 half-lives of the drug, whichever is longer, of entry into this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-12; Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Earvin Liang, Study Director — Bonti, Inc.
Locations (2):
- United States (2):
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Steve Yoelin, MD Medical Associates, INC., Newport Beach, California

REFERENCES:
- [Derived] Yoelin SG, Dhawan SS, Vitarella D, Ahmad W, Hasan F, Abushakra S. Safety and Efficacy of EB-001, a Novel Type E Botulinum Toxin, in Subjects with Glabellar Frown Lines: Results of a Phase 2, Randomized, Placebo-Controlled, Ascending-Dose Study. Plast Reconstr Surg. 2018 Dec;142(6):847e-855e. doi: 10.1097/PRS.0000000000005029. PMID 30489516

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Injection of placebo into five (5) 0.1 mL IM injections into glabellar area.
  Placebo injection
- EB-001 Dose 1 (1X): Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
  EB-001 injection
- EB-001 Dose 2 (3X): Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
  EB-001 injection 3X Dose 1
- EB-001 Dose 3 (9X): Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
  EB-001 injection 9X dose 1
- EB-001 Dose 4 (12X): Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
  EB-001 injection 12X Dose 1
- EB-001 Dose 5 (16X): Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
  EB-001 injection 16X Dose 1
- EB-001 Dose 6 (21X): Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
  EB-001 injection 21X Dose 1
- EB-001 Dose 7 (28X): Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
  EB-001 injection 28X Dose 1
Period: Overall Study
Arm/Group | Placebo | EB-001 Dose 1 (1X) | EB-001 Dose 2 (3X) | EB-001 Dose 3 (9X) | EB-001 Dose 4 (12X) | EB-001 Dose 5 (16X) | EB-001 Dose 6 (21X) | EB-001 Dose 7 (28X)
Started | 7 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 7 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- EB-001 Dose 1: 1st Dose in escalation paradigm.
  Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 2: 2nd Dose in escalation paradigm.
  Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 3: 3rd Dose in escalation paradigm.
  Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 4: 4th Dose in escalation paradigm.
  Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 5: 5thDose in escalation paradigm.
  Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 6: 6th Dose in escalation paradigm.
  Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 7: 7th Dose in escalation paradigm.
  Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- Total: Total of all reporting groups
Arm/Group | Placebo | EB-001 Dose 1 | EB-001 Dose 2 | EB-001 Dose 3 | EB-001 Dose 4 | EB-001 Dose 5 | EB-001 Dose 6 | EB-001 Dose 7 | Total
Number analyzed (Participants) | 7 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (8.48) | 52.0 (5.43) | 39.4 (16.13) | 52.2 (9.36) | 50.8 (6.50) | 45.4 (11.39) | 53.2 (4.66) | 42.6 (10.26) | 47.9 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 5 | 4 | 5 | 5 | 5 | 38
  Male | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3
  White | 5 | 3 | 4 | 2 | 5 | 2 | 4 | 5 | 30
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 42

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Assessment of GL Severity at Maximum Frown Using the Facial Wrinkle Scale (FWS).
Description: Subjects Achieving a 2 Grade Response At Maximum Frown On Any Study Day By Dose using the Facial Wrinkle Scale (FWS)
  The FWS is a four-point scale that indicates severity of GL as follows: 0 = none, 1 = mild, 2 = moderate, or 3 = severe.
  Each scale is a four-point photonumeric scale based on photographs incorporating each aspect to be evaluated in a stepwise manner.
Time Frame: After single injection treatment up to 42 days
Population: mITT
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Single Injection of placebo into five (5) 0.1 mL IM injections into glabellar area.
  Placebo injection
- EB-001 Dose 1 (1X): 1st Dose in escalation paradigm.
  Single Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 2 (3X): 2nd dose in escalation paradigm, 3X Dose 1.
  Single Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 3 (9X): 3rd Dose in escalation paradigm, 9X Dose 1.
  Single Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 4 (12X): 4th Dose in escalation paradigm, 12X Dose 1.
  Single Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 5 (16X): 5th Dose in escalation paradigm, 16X Dose 1.
  Single Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 6 (21X): 6th Dose in escalation paradigm, 21X Dose 1.
  Single Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
- EB-001 Dose 7 (28X): 7th Dose in escalation paradigm, 28X Dose 1.
  Single Injection of active drug into five (5) 0.1 mL IM injections into glabellar area.
Arm/Group | Placebo | EB-001 Dose 1 (1X) | EB-001 Dose 2 (3X) | EB-001 Dose 3 (9X) | EB-001 Dose 4 (12X) | EB-001 Dose 5 (16X) | EB-001 Dose 6 (21X) | EB-001 Dose 7 (28X)
Number analyzed (Participants) | 7 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Participants | 1 | 0 | 0 | 2 | 3 | 2 | 4 | 4

ADVERSE EVENTS:
Time Frame: 42 Days
Arm/Group | Placebo | EB-001 Dose 1 (1X) | EB-001 Dose 2 (3X) | EB-001 Dose 3 (9X) | EB-001 Dose 4 (12X) | EB-001 Dose 5 (16X) | EB-001 Dose 6 (21X) | EB-001 Dose 7 (28X)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 1/5 | 1/5 | 0/5 | 1/5 | 0/5 | 1/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | EB-001 Dose 1 (1X) (N=5) | EB-001 Dose 2 (3X) (N=5) | EB-001 Dose 3 (9X) (N=5) | EB-001 Dose 4 (12X) (N=5) | EB-001 Dose 5 (16X) (N=5) | EB-001 Dose 6 (21X) (N=5) | EB-001 Dose 7 (28X) (N=5)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flu-like Symptoms (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT02939326/Prot_SAP_000.pdf